CLINICAL TRIAL: NCT00866398
Title: Economic Evaluation German Drug-Eluting Stent Registry
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: IKKF GmbH (Unknown); IHF Ludwigshafen (Unknown); Cordis Medizinische Apparate GmbH (Other); Boston Scientific Corporation (Industry)
Responsible Party: Stefan N Willich, MD, MPH, MBA, Charité - Universitätsmedizin Berlin
Other Study IDs: 008
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Coronary Heart Disease
Keywords: coronary heart disease; chd; stent
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 DES: Patients receiving drug-eluting stent
- 2 BMS: Patients receiving bare metal stent

SUMMARY:
Since the advent of coronary stents, in-stent restenosis has proven to be the major limitation of interventional cardiology, occurring in as many as 30% of patients. Drug-eluting stents are specifically designed to prevent the problem of in-stent restenosis. They consist of a selective anti-proliferative drug, sirolimus, a controlled-release polymer, and a closed-cell stent delivery platform. Upon placement, sirolimus elutes into the vessel wall and stops the process of neointimal hyperplasia, thereby significantly reducing the incidence of in-stent restenosis.

The study "Economic Evaluation of the German Drug-Eluting Stent Registry" examines the cost-effectiveness of drug-eluting stents compared to bare-metal stents (BMS) in patients with coronary stenosis. The goal of the study is to examine whether the guideline-supported implantation of SES, despite the higher initial cost, improves the quality and economic outcomes of the treatment of patients with coronary stenosis. Secondarily, the study evaluates patient quality of life, impairment of daily activities, and re-intervention rates.

ELIGIBILITY:
Inclusion Criteria:

* Indication for coronary stent implantation
* Additional inclusion criteria BMS cohort:

  * Acute Coronary Syndrome
  * Diabetes Mellitus
  * Previous Percutaneous Coronary Intervention/Coronary Artery Bypass Graft
  * 3-Vessel Disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with coronary heart disease, eligible for stent implantation.
Sampling Method: Non-Probability Sample
Enrollment: 3973 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Cost equivalence of drug-eluting coronary stents versus bare metal stents | 12 months

SECONDARY OUTCOMES:
MACCE | 12 months
Quality of life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan N Willich, Prof, MD, MPH, Study Director — Charité University Medical Center